CLINICAL TRIAL: NCT03008733
Title: Descriptive Analysis of Morphological Aspects of Nerve by Ultra-high Frequency Ultrasound (30-50MHZ) in Demyelinating Neuropathies: Inflammatory Demyelinating Polyneuropathy Chronic (IPDC), Neuropathy Multifocal Motor Block of Conducting (NMMBC) and Neuropathy With Antibody A MAG
Acronym: EchoNerf
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16-AOIP-02
Record Dates: First submitted 2016-11-09; First posted 2017-01-02 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Polyradiculoneuropathy, Chronic Inflammatory Demyelinating
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- NMMCB (Active Comparator): patient with Neuropathies with Motrices Multifocal Conduction Block
  Interventions: Other: Ultrasound UHF peripheral nerves; Other: Electro myography surface nerves
- PICD (Active Comparator): patient with Inflammatory demyelinating polyneuropathy Chronicle
  Interventions: Other: Ultrasound UHF peripheral nerves; Other: Electro myography surface nerves
- anti MAG (Active Comparator): patient with neuropathy antibody Anti-MAG
  Interventions: Other: Ultrasound UHF peripheral nerves; Other: Electro myography surface nerves
- healthy (Placebo Comparator): healthy patient
  Interventions: Other: Ultrasound UHF peripheral nerves; Other: Electro myography surface nerves

INTERVENTIONS:
Other: Ultrasound UHF peripheral nerves — Ultrasound UHF peripheral nerves
Other: Electro myography surface nerves — Electro myography surface nerves

SUMMARY:
The use of nerve ultrasound for the diagnosis and monitoring of neuromuscular diseases is a promising growing field (1). Non-invasive and painless, ultrasound provides additional data electroneuromyography (EMG), with a spatial resolution at least as good as MRI, while being easily accessible and inexpensive.The polyradiculoneuritis Inflammatory Demyelinating Chronicles (IPDC), Neuropathies Motrices in Multifocal Conduction Blocks (NMMBC) and neuropathy associated with anti-MAG antibodies are among the major chronic inflammatory neuropathies with an autoimmune etiology. The diagnosis of these pathologies is based on the clinic, diagnostic tests and EMG. The interest not only in the diagnosis, but also for monitoring these pathologies using ultrasound analysis nerves has been demonstrated recently in several studies. However the limited resolution of current ultrasound images do not allow detailed study of the internal structure of the nerves which could later help deepen knowledge in this innovative field and can better understand the pathophysiological mechanism of the evolution of these pathologies .

To do this, the investigators have available a UHF ultrasound in the ultrasound department of the Nice University Hospital Pasteur Hospital 2 The investigators realize a descriptive analysis study, pilot, mono-centric, multi and prospective on patients followed in the center with a diagnosis of IPDC, a NMMBC or neuropathy with anti-MAG antibodies and control subjects matched by age and sex. All the patients and controls in this study will receive a briefing and must sign an informed consent.

They realize an ultrasound study of the nerve, using an ultra high frequency ultrasound system that will allow the assessment of anatomical structures of nerve (size, structure, vascularisation and assessment booklets). Ultrasound data will, in a second stage, compared with the data obtained with the EMG and clinical scores obtained using clinical rating scales. 40 subjects will be included, divided into four subgroups: 10 subjects with a diagnosis of IPDC (1), 10 subjects with a diagnosis of NMMBC (2), 10 subjects with a diagnosis of neuropathy antibody-anti MAG (3) and 10 control subjects with no signs of neuropathy at the EMG examination.

DETAILED DESCRIPTION:
The use of nerve ultrasound for the diagnosis and monitoring of neuromuscular diseases is a promising growing field (1). Non-invasive and painless, ultrasound provides additional data electroneuromyography (EMG), with a spatial resolution at least as good as MRI, while being easily accessible and inexpensive.The polyradiculoneuritis Inflammatory Demyelinating Chronicles (IPDC), Neuropathies Motrices in Multifocal Conduction Blocks (NMMBC) and neuropathy associated with anti-MAG antibodies are among the major chronic inflammatory neuropathies with an autoimmune etiology. The diagnosis of these pathologies is based on the clinic, diagnostic tests and EMG. The interest not only in the diagnosis, but also for monitoring these pathologies using ultrasound analysis nerves has been demonstrated recently in several studies. However the limited resolution of current ultrasound images do not allow detailed study of the internal structure of the nerves which could later help deepen knowledge in this innovative field and can better understand the pathophysiological mechanism of the evolution of these pathologies .

To do this, the investigators have available a UHF ultrasound in the ultrasound department of the Nice University Hospital Pasteur Hospital 2 The investigators realize a descriptive analysis study, pilot, mono-centric, multi and prospective on patients followed in the center with a diagnosis of IPDC, a NMMBC or neuropathy with anti-MAG antibodies and control subjects matched by age and sex. All the patients and controls in this study will receive a briefing and must sign an informed consent.

They realize an ultrasound study of the nerve, using an ultra high frequency ultrasound system that will allow the assessment of anatomical structures of nerve (size, structure, vascularisation and assessment booklets). Ultrasound data will, in a second stage, compared with the data obtained with the EMG and clinical scores obtained using clinical rating scales. 40 subjects will be included, divided into four subgroups: 10 subjects with a diagnosis of IPDC (1), 10 subjects with a diagnosis of NMMBC (2), 10 subjects with a diagnosis of neuropathy antibody-anti MAG (3) and 10 control subjects with no signs of neuropathy at the EMG examination.

The main objective of this pilot study is to provide a descriptive analysis of the morphology of the nerves with an ultra high frequency ultrasound in subgroups of CIDP patients, anti-MAG antibodies and neuropathy NMMBC and controls. The thickness of the epineurium, the hallmarks of fascicular organization, Doppler vascularity, the nerve-sectional area, the specification of the section surface, nerve hypertrophy, the thickness of the perineurium and ultrastructural characterization of the different fascicular organization typologies will be well analyzed in order to better understand the specific sonographic characteristics of each disease compared with controls, no data exist at present in the literature with such image resolution.

Secondary objectives:

1. Compare the morphological characteristics obtained by ultra high frequency ultrasound between different subjects subgroups according to the morphological data collected and sonographic scores: evaluation of nerve hypertrophy (intra- and inter-ratio nerve nerve) (4 ) and intra-fascicular nerve and nerve cross-ratio.
2. To study the correlation between sonographic and clinical scores scores in different subjects subgroups using functional assessment scales: MRC score, R-ODS score, INCAT, ONLS, ataxia Score and a torque rating of grip strength.
3. To study the correlation between sonographic scores and electrophysiological scores by making a électroneurogramme (ENG) in the different subjects of subgroups: the amplitude and distal motor latency for distal motor conduction, the motor conduction velocities, the presence of time dispersion or of a conduction block to the stepped motor conduction, the latency of the waveform F to the proximal motor conduction and the amplitude of the sensory potential for sensory conduction.

ELIGIBILITY:
Inclusion Criteria:

common inclusion criteria for all subjects:

* Man or woman age ≥ 18 years.
* Affiliation to social security.
* Signature of informed consent.

Inclusion criteria for CIDP patients:

- Patients with certain IPDC according to the following criteria defined by the EFNS 2010:

At least one of demyelination following criteria must be present:

* Extension of the Distal Motor Latency ≥ 50% above the limit Normale Supérieure (LNS) in 2 nerves (excluding impairment of the median nerve at the wrist due to carpal tunnel syndrome);
* Reducing the speed of conduction Average ≥ 30% below the normal limit Lower (LNI) in 2 nerves;
* Extension of the latency of the F wave ≥ 30% above the ULN in two nerves (≥ 50% of the LNS if the amplitude of distal negative peak PAGM (Action Potential Global Muscle) is < 80% of the LNI;
* Lack wave F in 2 nerves if these nerves have an amplitude of the negative peak of the distal PAGM ≥ 20% of the LNS + ≥ 1 other parameter of demyelination in * ≥ 1 other nerve;
* Conduction Block partial engine: decreased range ≥ 50% of the negative peak of the proximal to the distal PAGM PAGM, if the negative peak of the distal PAGM ≥ 20% LNI in 2 nerves or nerve + 1 ≥ 1 another parameter of demyelination in ≥ 1 * other nerve;
* abnormal temporal dispersion (> 30% increase in duration between the negative peak of the proximal and distal PAGM) ≥ 2 in nerves;
* PAGM distal length (interval between the start of the negative peak and its return to baseline) in ≥ 1 nerve (median ≥ 6.6 ms, ulnar ≥ 6.7 ms ≥ 7.6 ms peroneal, tibial ≥ 8.8 ms) + 1 ≥ another parameter * demyelination in ≥ 1 other nerve.

Inclusion criteria for patients NMMBC:

* Patients with certain NMMBC according to the following criteria defined by the EFNS (2010):

  * Weak slowly progressive or progressive members in spurts, and focal asymmetric, due to damage of the driving motor nerve distribution in at least two nerves, for over a month.
  * Lack of objective sensory abnormality except for sensory anomalies minor vibrations in the lower limbs.
  * In a nerve:
* conduction block some engine.
* Conduction normal sensory nerves in the segments of the upper limbs with conduction block.

  * No evidence of upper motor neuron.
  * Lack of significant bulbar weakness.
  * Sensory impairment less marked than the minor loss of sensitivity to vibrations in the lower limbs.
  * symmetrical weakness Lack broadcasts during the first weeks.

Inclusion criteria for the neuropathy patients with anti-MAG antibody:

- Patients with neuropathy with anti-MAG antibody according to criteria defined by the EFNS (2010):

* electrophysiological criteria:

  * symmetrical uniform reduction of conduction velocity; more severe at that sensory motor.
  * Distal Motor Latency disproportionately long: Index of Distal Latency ≤ 0.25.
  * Potential sural missing.
* Clinical criteria:

  * Early disease> 50 years.
  * ataxia associated with shaky hands.
* Biological criteria:

  * IgM monoclonal rate lower than 10 g / l, or greater than 10 g / l in the context of Waldenström's macroglobulinemia.
  * Presence of anti-MAG antibody (Myelin-Associated Glycoprotein).

Exclusion Criteria:

* Presence of risk factors associated neuropathic disease (diabetes, chronic alcoholism, kidney failure, HIV status, Lyme disease, vasculitis or any other factor which, in the judgment of the investigator, could pose a risk).
* A patient pathology judged by the investigator as interfering with the proper conduct of the study.
* Positive pregnancy test. A urine pregnancy test will be performed for women of childbearing age. Results will be communicated to the patient by a doctor of his choice.
* Refusal of the subject to participate in the study.
* Topic guardianship or curatorship.
* Inability of the subject to cooperate.
* No affiliation to a social security scheme (beneficiary or assignee).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
morphology of the nerves by means of an ultra-high frequency ultrasound in patients subgroups CIDP, anti-MAG antibodies and NMMBC neuropathy and control subjects. | through study completion an average of 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No